CLINICAL TRIAL: NCT00854490
Title: Follow-up Study of Small-intestinal Mucosal Injuries in Chronic Non-steroidal Anti-inflammatory Drugs (NSAIDs)-Users
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nagoya University (Other)
Responsible Party: Naoki Ohmiya, Department of Gastroenterology, Nagoya University Hospital
Other Study IDs: NO-002
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Enteropathy
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to evaluate the long-term clinical significance of small-intestinal mucosal injuries in chronic NSAIDs-users.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* 20 to 85 years of age
* RA, OA, or low back pain
* taking oral diclofenac sodium over 3 months
* No change of drugs before 3 months
* under 5 mg of corticosteroid use
* CRP < 1mg/dl

Exclusion Criteria:

* known or suspected small-bowel disease, including Crohn's disease and seronegative arthritis
* prostaglandins, metronidazole or salazosulfapyridine
* can not swallow
* with pacemaker
* after gastrointestinal operation
* serious concomitant cardiovascular, endocrine, gastrointestinal(including symptoms of ileus), neurologic, psychiatric, renal, or respiratory disease.
* any other conditions that the investigator feels would interfere with data interpretation or create under risk

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic NSAID users
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-10

CONTACTS AND LOCATIONS:
Locations (1):
- Nagoya University Hospital, Nagoya, Aichi-ken, Japan